CLINICAL TRIAL: NCT02105870
Title: A Randomized Control Trial of Intracoronary Reopro to Improve Coronary Microvascular Function
Brief Title: A Randomized Trial of Intracoronary Reopro to Improve Coronary Microvascular Function
Acronym: Intracor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, A/P Andrew Wilson, Associate Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVH 001
Record Dates: First submitted 2013-12-09; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracoronary abciximab (Reopro) (Experimental): Intracoronary abciximab (Reopro)
  Interventions: Drug: Abciximab
- Control group (Placebo Comparator): Intracoronary Reopro

INTERVENTIONS:
Drug: Abciximab — This drug will be administered intracoronary before percutaneous coronary intervention.
  Other Names: Reopro
  Arms: Intracoronary abciximab (Reopro)

SUMMARY:
Microvascular dysfunction is a key determinant of pathogenesis and outcome in patients suffering an acute myocardial infarction.

The investigators hypothesise that treatment with intracoronary abciximab, a potent anti platelet agent, at the time of coronary stent insertion, will improve microvascular function.

DETAILED DESCRIPTION:
The index of microcirculatory resistance (IMR), an invasive measure of coronary microvascular function, correlates with clinical outcomes in patients with stable angina and ST elevation myocardial infarction. The glycoprotein IIb/IIIa receptor inhibitor, abciximab, improves coronary microvascular function and reduces major cardiac adverse events in patients with acute coronary syndromes. This study will investigate whether an intracoronary bolus of abciximab in patients with non-ST elevation myocardial infarction decreases IMR and improves microvascular function.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute coronary syndromes

Exclusion Criteria:

* Patient with untreated malignancy, disseminated malignancy, active inflammatory diseases, active infectious diseases patients unable to give informed consent Patients with STEMI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Index of Microvascular Resistance | within 3 hours
  We will assess IMR in the catheterisation laboratory immediately before PCI, then intracoronary reopro or placebo will be administered and we will re-assess IMR 15 minutes post delivery of the study drug. Finally we will perform PCI and immediately measure IMR post-procedure.

SECONDARY OUTCOMES:
Incidence of periprocedural myocardial infarction | within 24 hours
  We will assess for periprocedural myocardial infarction 8 to 24 hours post PCI

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilson, MD PhD, Principal Investigator — University of Melbourne
Locations (1):
- St Vincent's Hospital, Fitzroy, Victoria, Australia